CLINICAL TRIAL: NCT04592003
Title: French Colorectal ESD Cohort in Experts Centers
Acronym: FECCo
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20-0021_FECCo
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer Colorectal; Polyps Colorectal; Endoscopic Submucosal Resection
Keywords: Cancer colorectal; Polyps colorectal; Endoscopic submucosal resection
MeSH Terms: conditions — Colonic Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FECCo : French Esd Colorectal Cohort in Experts Centers: All patients over 18 years of age referred for submucosal dissection of a polyp or a colorectal LST in the French centers participating in the cohort.
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — Endoscopic submucosal dissection

SUMMARY:
Initially developed in Japan for the treatment of endemic superficial gastric cancers, endoscopic submucosal dissection (ESD) allows resection of pre-neoplastic and neoplastic lesions of the digestive tract into a single fragment. It allows a perfect pathological analysis, and decreases the rate of recurrence of the adenoma to less than 2%. However, this procedure, which is technically more challenging, is also more risky (perforation rate at 4% vs. 1% for WF-EMR) and longer. Submucosal dissection is also more expensive in terms of equipment, but this difference can be offset by the cost of the high number of iterative colonoscopies required in patients who have had endoscopic resection by WF-EMR.

Scientific debate is agitating the Western world1,2 and Japanese experts do not perform WF-EMR anymore, whereas no comparative prospective study has compared these two procedures.

A lot of centers in France performed colorectal ESD even for benign lesions and nationwide data about safety and efficiency is required to confirm the place of ESD for treatment of large superficial colorectal lesions.

The aim of this French multicenter cohort is to analyze the results of colorectal submucosal dissection on a large scale.

DETAILED DESCRIPTION:
Initially developed in Japan for the treatment of endemic superficial gastric cancers, endoscopic submucosal dissection (ESD) allows resection of pre-neoplastic and neoplastic lesions of the digestive tract into a single fragment. It allows a perfect pathological analysis, and decreases the rate of recurrence of the adenoma to less than 2%. However, this procedure, which is technically more challenging, is also more risky (perforation rate at 4% vs. 1% for WF-EMR) and longer. Submucosal dissection is also more expensive in terms of equipment, but this difference can be offset by the cost of the high number of iterative colonoscopies required in patients who have had endoscopic resection by WF-EMR.

Scientific debate is agitating the Western world1,2 and Japanese experts do not perform WF-EMR anymore, whereas no comparative prospective study has compared these two procedures.

A lot of centers in France performed colorectal ESD even for benign lesions and nationwide data about safety and efficiency is required to confirm the place of ESD for treatment of large superficial colorectal lesions.

The aim of this French multicenter cohort is to analyze the results of colorectal submucosal dissection on a large scale.

ELIGIBILITY:
Inclusion Criteria:

All patients addressed for a colorectal ESD

Exclusion Criteria:

Opposition notified in the context of a non-opposition form after reading the information notice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients addressed for a colorectal ESD
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
R0 Resection rate of submucosal dissection for superficial colorectal lesions | Month 1
  R0 Resection rate according to the definition of of the European Society of Gastrointestinal Endoscopy.

SECONDARY OUTCOMES:
Endoscopic recurrence rate during the first endoscopic follow-up | Month 6
  Recurrence during the first endoscopic follow-up will be defined by the presence of adenoma or adenocarcinoma at the resection scar, whether visible or not, and confirmed by systematic biopsies of the resection scar.
Monobloc resection rate | Day 1
  Monobloc resection is defined as resection of the lesion in a single piece.
Monobloc resection rate exclusively in ESD. | Day 1
  Monobloc resection exclusively by ESD is defined as resection of the lesion in a single piece using submucosal dissection only, without the use of a diathermic loop (hybrid technique).
Curative resection rate | Month 1
  Curative resection is defined according to the recommendations of the European Society of Digestive Endoscopy as a monobloc R0 dissection without any negative anatomopathological criteria (well-differentiated lesion, no emboli, no budding > 1, submucosal infiltration < 1 mm).
Optimal dissection rate | Month 1
  Optimal dissection is defined as exclusive R0 dissection without perforation, with a resection speed > 20 mm2/min.
30-day complication rate | Month 1
  * Per-procedural perforation: breach of the colonic musculature with visualization of the peritoneal cavity.
  * Post-procedural perforation (≤ 30 days): abdominal pain associated with fever or inflammatory syndrome and presence of extraluminal air on abdominal-pelvic CT scan, in the absence of per-procedural perforation.
  * Per-procedural hemorrhage: considered a complication only if it leads to interruption of the procedure.
  * Post-procedural hemorrhage: rectal bleeding or melena requiring hospitalization (or prolonged hospitalization) or endoscopic hemostasis.
Curative endoscopic resection rate without surgical management at 36 months | Month 36
  Curative endoscopic resection without surgery is defined by the absence of adenoma or adenocarcinoma at the resection scar after 36 months of follow-up, regardless of the number of endoscopic treatments required.
Number of metachronous colorectal lesions at 36 months | Month 36
  A metachronous lesion is defined as the presence of a new superficial colorectal lesion during one of the endoscopic checks, a lesion not visualized during one of the previous examinations.
Surgery rate at 36 months | Month 36
  Any colorectal surgery will be taken into account, whether due to failure of the endoscopic procedure, recurrence, a complication of the procedure, or an anatomopathological reason.
Recurrence rate at 36 months | Month 36
  Recurrence at 36 months will be defined by the presence of adenoma or adenocarcinoma at the resection scar, whether visible or not, and confirmed by systematic biopsies of the resection scar.
Effectiveness of histological prediction of superficial colorectal lesions treated according to the technological tools used. | Month 1
  The histological prediction of resected lesions will be established using validated classifications (Paris, SANO, NICE, KUDO, JNET, CONECTT). It will be compared with the definitive histological results to assess their sensitivity, specificity, and diagnostic accuracy within the cohort.
Impact of center volume on oncological outcomes, technical outcomes, and procedural complications. | Month 1
  Oncological, technical, and complication outcomes will be analyzed according to the annual volume of the centers (low volume = < 50 ESDs per year; intermediate volume = between 50 and 100 procedures per year; high volume = > 100 procedures per year).
Compare oncological and technical outcomes and procedural complications based on colonic or rectal location. | Month 1
  Oncological, technical, and complication outcomes will be analyzed according to the colonic or rectal location of the lesion.
Compare procedural outcomes based on the different traction strategies used | Month 1
  Oncological, technical, and complication outcomes will be analyzed according to the traction system used for the procedure, matching lesions according to difficulty criteria validated by the literature.
Analyze the learning curve of new trainees at the time of implementation of the submucosal dissection curriculum of the French Society of Digestive Endoscopy. | statitistic analysis
  The learning curve of trainees will be used to evaluate oncological, technical, and complication outcomes using the LC CUSUM method.
Creation of a difficulty score predicting the success of ESD (R0 resection without perforation) | Month 1
  A difficulty score predicting success (R0 without perforation) will be created by performing a multivariate analysis according to the TRIPOD GUIDELINES using a derivation cohort and validated on a derivation cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Jacques, Pr, Principal Investigator — Service d'Hépato-Gastro-Entérologie et Nutrition du CHU de LIMOGES
Locations (25):
- France (25):
  - CHU d'Amiens, Amiens
  - Clinique de l'Anjou, Angers
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - CHU de Dijon, Dijon
  - CHU de Limoges, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hôpital Jean Mermoz, Lyon
  - Hôpital Européen, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - Clinique Jules Vernes, Nantes
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - Hôpital St Antoine, Paris
  - Hôpital Cochin - APHP, Paris
  - Hôpital St Joseph, Paris
  - Hôpital Européen Georges Pompidou-APHP, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - Clinique Santé Atlantique, Saint-Herblain
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Van der Voort V, Schaefer M, Wallenhorst T, Lepilliez V, Degand T, Le Baleur Y, Leclercq P, Berger A, Chabrun E, Brieau B, Barret M, Rahmi G, Legros R, Rivory J, Leblanc S, Vanbiervliet G, Alfarone L, Magne J, Zeevaert JB, Albouys J, Perrod G, Yzet C, Lepetit H, Belle A, Chaussade S, Rostain F, Dahan M, Lupu A, Chevaux JB, Pioche M, Jacques J; FECCo Group collaborators. Rectal versus colonic submucosal cancer rates and procedural outcomes in large non-pedunculated polyps: French ESD registry data. Gut. 2025 Oct 12:gutjnl-2024-332970. doi: 10.1136/gutjnl-2024-332970. Online ahead of print. PMID 41083216
- [Derived] Yzet C, Wallenhorst T, Jacques J, Figueiredo Ferreira M, Rivory J, Rostain F, Masgnaux LJ, Grimaldi J, Legros R, Lafeuille P, Albouys J, Subtil F, Schaefer M, Pioche M. Traction-assisted endoscopic submucosal dissection for resection of ileocecal valve neoplasia: a French retrospective multicenter case series. Endoscopy. 2024 Oct;56(10):790-796. doi: 10.1055/a-2316-4910. Epub 2024 Apr 29. PMID 38684193
- [Derived] Yzet C, Le Baleur Y, Albouys J, Jacques J, Doumbe-Mandengue P, Barret M, Abou Ali E, Schaefer M, Chevaux JB, Leblanc S, Lepillez V, Privat J, Degand T, Wallenhorst T, Rivory J, Chaput U, Berger A, Aziz K, Rahmi G, Coron E, Kull E, Caillo L, Vanbiervliet G, Koch S, Subtil F, Pioche M. Use of endoscopic submucosal dissection or full-thickness resection device to treat residual colorectal neoplasia after endoscopic resection: a multicenter historical cohort study. Endoscopy. 2023 Nov;55(11):1002-1009. doi: 10.1055/a-2116-9930. Epub 2023 Jul 27. PMID 37500072
- [Derived] Patenotte A, Yzet C, Wallenhorst T, Subtil F, Leblanc S, Schaefer M, Walter T, Lambin T, Fenouil T, Lafeuille P, Chevaux JB, Legros R, Rostain F, Rivory J, Jacques J, Lepilliez V, Pioche M. Diagnostic endoscopic submucosal dissection for colorectal lesions with suspected deep invasion. Endoscopy. 2023 Feb;55(2):192-197. doi: 10.1055/a-1866-8080. Epub 2022 Jun 1. PMID 35649429